CLINICAL TRIAL: NCT01189578
Title: Neural Correlates of Craving and Impulsivity in Recreational Cocaine Users
Brief Title: Brain Imaging of Cocaine Craving in Recreational Cocaine Users
Status: Completed | Type: Observational
Sponsor: James J. Prisciandaro (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, James J. Prisciandaro, Assistant Professor, Medical University of South Carolina
Organization: Medical University of South Carolina (Other)
Other Study IDs: HR# 20276; R01DA023188 (NIH)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Cocaine Related Disorders
Keywords: Recreational; cocaine; fMRI; neuroimaging; craving; impulsivity
MeSH Terms: conditions — Cocaine-Related Disorders; Impulsive Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Recreational cocaine users: Individuals who have used cocaine in the past 3 months, but do not meet DSM-IV-TR diagnostic criteria for Cocaine Dependence.

SUMMARY:
The purpose of this study is to compare individuals with cocaine dependence to recreational users of cocaine in terms of their brain reactivity to cocaine cues, in hopes that this comparison may help us better understand the transition from recreational to compulsive cocaine use.

DETAILED DESCRIPTION:
Chronic cocaine exposure is associated with an intensified and broadened pattern of neural reactivity to cocaine and cocaine cues; prolonged use is also associated with prefrontal abnormalities during response inhibition. Limited research suggests that recreational cocaine use has similar, but attenuated, effects on neural functioning. Unfortunately, very little research has directly compared cocaine dependent individuals and recreational cocaine users in terms of their neural reactivity to cocaine cues and response inhibition. Such comparisons could help to elucidate the pathological neuroplasticity associated with the transition from cocaine use to dependence. The proposed study will assess neural reactivity to cocaine cues and response inhibition in recreational cocaine users using fMRI. These data will be compared to data from the baseline visit of an ongoing IRB approved investigation (NCT00759473) in cocaine dependent individuals that is using the same experimental procedures as the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
* Subjects must report having used cocaine within the past 3 months. Subjects may meet criteria for abuse, but not dependence on any other substance with the exception of nicotine, marijuana and alcohol.
* Use of one of the following methods of birth control by female subjects: birth control pills, barrier methods (diaphragm or condoms with spermicide or both), surgical sterilization, use of an intra-uterine contraceptive device, or complete abstinence from sexual intercourse.
* Subjects must live within a 50-mile radius of the research facility and have reliable transportation.
* Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) prior to the experiment.
* Subjects must be right-handed.

Exclusion Criteria:

* Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
* Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect heart rate or skin conductance measurement.
* Subjects with a history of or current psychotic disorder as this may impact cue reactivity.
* Subjects who are unwilling or unable to maintain abstinence from alcohol and other drugs of abuse (except nicotine).
* Subjects meeting DSM-IV criteria for substance dependence (other than nicotine, marijuana, or alcohol) within the past 60 days. Subjects may not meet criteria for cocaine dependence at any time.
* Subjects currently taking B-blockers, anti-arrhythmic agents, psychostimulants or any other agents known to interfere with heart rate and skin conductance monitoring.
* Subjects with a history of epilepsy or seizure disorder.
* Subjects with significant liver impairment.
* The need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications which could potentially interfere with fMRI.
* Clinically significant psychiatric or medical problems that would impair participation or limit ability to participate in scan.
* Persons with ferrous metal implants or pacemaker since fMRI will be used.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen T Brady, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States